CLINICAL TRIAL: NCT03237663
Title: Safety of An Oral O1 / O139 Cholera Vaccine (Enteric Capsules) Through Phase I Clinical Trial in China
Brief Title: Safety of An Oral O1 / O139 Cholera Vaccine (Enteric Capsules)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT023
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Safety of the Oral O1 / O139 Cholera Vaccine (Enteric Capsules)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One enteric capsule (Experimental)
  Interventions: Biological: The oral O1 / O139 cholera vaccine (enteric capsules)
- Two enteric capsule (Experimental)
  Interventions: Biological: The oral O1 / O139 cholera vaccine (enteric capsules)

INTERVENTIONS:
Biological: The oral O1 / O139 cholera vaccine (enteric capsules)

SUMMARY:
Cholera is an acute enteric infectious disease caused by the bacterium Vibrio cholera, leading to watery diarrhea and loss of fluids from the small intestines. The World Health Organization (WHO) estimates that up to 4.3 million cholera cases annually with more than 100,000 of them result in death in worldwide. Cholera is mainly caused by the O1 or O139 serogroups of V. cholera. Vaccination has been shown to be a cost-effective, more immediate option for cholera control and prevention. Injectable vaccine is not recommended by the World Health Organization (WHO) mainly because of its limited efficacy and short duration of protection. However, the inactivated whole-cell, bivalent O1 and O139 cholera vaccine have provided evidence of substantial protective efficacy. With the goal of making an ideal low-cost OCV that could be used in cholera-endemic countries, a phase I trial was conducted to estimate safety of the oral O1 / O139 cholera vaccine (enteric capsules).

DETAILED DESCRIPTION:
Cholera is an acute enteric infectious disease caused by the bacterium Vibrio cholera, leading to watery diarrhea and loss of fluids from the small intestines. The disease can quickly lead to severe dehydration and death without proper and timely management. The World Health Organization (WHO) estimates that up to 4.3 million cholera cases annually with more than 100,000 of them result in death in worldwide. The high morbidity and consequent mortality caused by cholera is attributable to several factors, including lack of access to safe drinking water, poor sanitation and poor hygiene practices and transmitted via the fecal-oral route by ingesting food or water contaminated with the bacterium. Cholera is a significant public health issue in many developing countries in Africa, Southeast Asia, the Caribbean, and South America, and is rare in industrial countries with most cases occurring in travelers who have visited cholera-affected areas.

Cholera is mainly caused by the O1 or O139 serogroups of V. cholerae among the more than 200 V. cholerae serogroups, O1 strains are divided into two biotypes: Classical and El Tor. Each biotype can be further divided into 3 serotypes: Inaba, Ogawa, Hikojima. V. cholerae O1 has been shown to be responsible for the first six cholera pandemics. In 1992, a new V. cholerae serogroup O139 emerged and it has caused epidemics that spanned most of Asia. This strain was a genetic derivative of El Tor biotype in which the O1 biosynthetic genes were replaced by the O139 biosynthetic genes. Both V. cholerae O1 and O139 can produce an enterotoxin, which causes serious diarrhea, causing dehydration, and can lead to death in a few days.

Vaccination has been shown to be a cost-effective, more immediate option for cholera control and prevention. Injectable vaccine is not recommended by the World Health Organization (WHO) mainly because of its limited efficacy less than 50% and short duration of protection almost no more than six months. Enteric vaccination has already been regarded as the most effective approach to control such illnesses as well as to prevent cholera in endemic countries. The inactivated whole-cell, bivalent O1 and O139 cholera vaccine have provided evidence of substantial protective efficacy up to 60% at least 3-5 years. In 2011 the first low-cost oral cholera vaccine for international use was given prequalification by the World Health Organization (WHO). With the goal of making an ideal low-cost OCV that could be used in cholera-endemic countries, a phase I trial was conducted to estimate safety of the oral O1 / O139 cholera vaccine (enteric capsules), in order to fulfill the requirements of WHO. On the other hand, China is a non-endemic country of cholera, it will also can provided a safe and convenient vaccine for the travellers who visited cholera-affected areas.

ELIGIBILITY:
Inclusion Criteria:

* - Healthy adults aged 16-60 years old as established by medical history and clinical examination.
* The subjects' guardians are able to understand and sign the informed consent.
* Subjects who can and will comply with the requirements of the protocol.
* Hemoglobin: 110-150g/L (female), 120-160g/L (male)
* Leukocyte count: 4.0-10.0×109 /L
* Lymphocyte count: 0.8-4.5×109 /L
* Platelet count: 100-300×109/L
* Alanine aminotransferase: (ALT)0-40U/L
* Serum creatinine: 44-106μmol/L
* Subjects with temperature ≤37.0°C on axillary setting.

Exclusion Criteria:

* Pregnant or lactating women;
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine.
* Have serious side effects to vaccine, such as allergies, hives, breathing difficulties, angioneurotic oedema or abdominal pain;
* abdominal pain or diarrhea;
* asthma, in the past two years, unsteady and require emergency treatment, hospitalization, intubation, oral administration or intravenous corticosteroids;
* Diabetes (type I or II), not including gestational diabetes;
* Thyroid disease
* Serious angioneurotic edema in the past three years, or in need of treatment in the past 2 years
* Hypertension, over 145/95 mmHg
* Blood coagulation disorder (such as the lack of clotting factors, clotting hemorrhagic disease, abnormal platelet) or apparent bruises or blood coagulation disorder
* Malignant tumor, activity or have been treated tumor without cure or may relapse during the test;
* Epilepsy, not including fever epilepsy under 2 years old or alcoholic epilepsy in the first 3 years after temperance or idiopathic epilepsy in the past three years and do not need treatment;
* No spleen, functional asplenia, and any situation caused by no spleen or splenectomy;
* Guillain-Barre syndrome
* Pregnancy test positive women
* Any prior administration of immunodepressant or corticosteroids, and antianaphylactic treatment, cytotoxic therapy in last 6 months.
* Any prior administration of blood products in last 3 month.
* Any prior administration of other research medicines in last 1 month.
* Any prior administration of attenuated live vaccine in last 1 month.
* Any prior administration of subunit or inactivated vaccines in last 2 weeks.
* Had fever before vaccination, subjects with temperature >37.0°C on axillary setting.
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives.

Exclusion Criteria for the second and third dose:

* Subject who must be excluded according to the exclusion criteria for the last dose
* Any serious adverse events caused by vaccination.
* Adverse reactions no less than grade 3 within 72 hours after the last vaccination .

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2016-11-05 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects reporting solicited adverse reactions. | Day 7 post-each dose
  Proportion of subjects reporting adverse reactions on day 7 post-each dose.

SECONDARY OUTCOMES:
Proportion of subjects reporting unsolicited adverse events. | Day 28 post-each dose.
  Proportion of subjects reporting unsolicited adverse events on day 28 post-each dose.